CLINICAL TRIAL: NCT06595251
Title: Community Park-Based Programs for Health Promotion: Fit2Play Prospective Cohort Study
Acronym: F2P
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Miami-Dade County Parks and Recreation (Other); The Children's Trust, Miami FL (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105669
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Obesity; Hypertension; Prehypertension; Anxiety; Well-being; Depression; Low Physical Fitness; Psychological
Keywords: Youth; Afterschool; Parks and Recreation; Mental Health; Physical Health; Physical Activity; Exercise
MeSH Terms: conditions — Overweight; Obesity; Hypertension; Prehypertension; Anxiety Disorders; Depression; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fit2Play Program
  Interventions: Other: Fit2Play curriculum

INTERVENTIONS:
Other: Fit2Play curriculum — Fit2Play is a daily after-school park-based program (Monday-Friday, 2 PM-6 PM) that comprises (1) 60 minutes of physical activity that incorporates multiple sports (soccer, kickball, flag football) and activities from Sports, Play and Active Recreation for Kids (SPARK), a play- and evidenced-based, outcome-oriented, structured, active recreation program for children with a focus on developing and improving motor skills, movement knowledge, social and personal skills; and (2) 20-30 minutes of nutrition education lessons 1-2 times per week that incorporate EmpowerMe4Life, a health and wellness curriculum aligned to the National Health Education Standards for fifth grade and grounded in the American Heart Association's scientific recommendations in promoting heart-healthy lifestyles. Miami-Dade Parks and Recreation is the sponsor of the Fit2Play prospective cohort study. Duke is conducting a secondary data analysis on data collected as part of the Fit2Play study.

SUMMARY:
The Fit2Play prospective cohort study examines the effects of a park-based youth physical activity afterschool program on youth participant fitness and mental health outcomes. Duke will perform a secondary analysis of the data collected as part of the Fit2Play prospective cohort study run by Miami-Dade County Parks and Recreation.

DETAILED DESCRIPTION:
The Fit2Play prospective cohort study examines the effects of a park-based youth physical activity afterschool program on youth participant fitness and mental health outcomes. The Fit2Play program was designed by a team of MDPROS professionals and UM faculty. It is a daily after-school park-based program (Monday-Friday, 2 PM-6 PM) that comprises (1) 60 minutes of physical activity that incorporates multiple sports (soccer, kickball, flag football) and activities from Sports, Play and Active Recreation for Kids (SPARK), a play- and evidenced-based, outcome-oriented, structured, active recreation program for children with a focus on developing and improving motor skills, movement knowledge, social and personal skills; and (2) 20-30 minutes of nutrition education lessons 1-2 times per week that incorporate EmpowerMe4Life, a health and wellness curriculum aligned to the National Health Education Standards for fifth grade and grounded in the American Heart Association's scientific recommendations in promoting heart-healthy lifestyles. Fit2Play programming is implemented by park coaches, who are hired with health and wellness training and/or education-specific background(s) with at least a high school degree. Participants are divided into younger (6-9 years) and older (10-14 years) age groups regardless of weight status, and coaches choose daily age-appropriate SPARK and other physical activities for each group. With an oversight from a registered dietician, similarly, the UM-MDPROS team has expanded the EmpowerMe4Life curriculum to include younger (6-9 years) and older (10-14 years) age group modules.

The research team includes a large community organization (Miami-Dade County Parks and Recreation Department). All consented Fit2Play participants (400-800 per year) complete a baseline (August/September) and post-test (May/June) assessment during each school year of participation that include demographic, mental health symptom questionnaires, satisfaction surveys, and on-site physical fitness and biometric measurements. Data collection is performed by a core MDPROS measurement team who are trained and certified by University of Miami School of Medicine faculty. In addition, MDPROS bachelor/master's level recreation directors oversee on-site measurement procedures and collection of all predata and postdata to ensure measurement fidelity. Data are then uploaded to a shared (parks and university) database via a data management team.

ELIGIBILITY:
Inclusion Criteria:

* All participants enrolled in the Miami-Dade Fit2Play study will be included in this secondary analysis

Exclusion Criteria:

* Anyone not enrolled in the Miami-Dade Fit2Play study will be excluded from this secondary analysis

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fit2Play aims to enroll youth ages 6-14 years who are majority Hispanic and non-Hispanic black, 50% male; approximately 60% of the population will be normal weight, 15% with overweight, and 25% with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 12-72 MONTHS
Change in Height | Baseline, 12-72 MONTHS
Change in Waist-to-Hip Circumference | Baseline, 12-72 MONTHS
Change in Pulse | Baseline, 12-72 MONTHS
Change in Blood Pressure | Baseline, 12-72 MONTHS
Change in PACER score | Baseline, 12-72 MONTHS
Change in sit-and-reach test | Baseline, 12-72 MONTHS
Change in number of push-ups | Baseline, 12-72 MONTHS
Change in number of sit-ups | Baseline, 12-72 MONTHS
Change in Kidscreen-27 | Baseline, 12-72 MONTHS
Change in GAD-7 | Baseline, 12-72 MONTHS
Change in PHQ-8 | Baseline, 12-72 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'Agostino, DPH, MS, MEd, MA, Principal Investigator — Duke University
Locations (1):
- Miami-Dade County Parks, Recreation and Open Spaces Department, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Agostino EM, Patel HH, Hansen E, Mathew MS, Nardi M, Messiah SE. Longitudinal analysis of cardiovascular disease risk profile in neighbourhood poverty subgroups: 5-year results from an afterschool fitness programme in the USA. J Epidemiol Community Health. 2018 Mar;72(3):193-201. doi: 10.1136/jech-2017-209333. Epub 2017 Nov 24. PMID 29175865
- [Background] Booth JV, Messiah SE, Hansen E, Nardi MI, Hawver E, Patel HH, Kling H, Okeke D, D'Agostino EM. Objective Measurement of Physical Activity Attributed to a Park-Based Afterschool Program. J Phys Act Health. 2021 Mar 1;18(3):329-336. doi: 10.1123/jpah.2020-0162. Epub 2021 Jan 31. PMID 33524953
- [Background] D'Agostino EM, Patel HH, Hansen E, Mathew MS, Nardi MI, Messiah SE. Effect of participation in a park-based afterschool program on cardiovascular disease risk among severely obese youth. Public Health. 2018 Jun;159:137-143. doi: 10.1016/j.puhe.2018.02.025. Epub 2018 Mar 27. PMID 29599055
- [Background] Messiah SE, D'Agostino EM, Hansen E, Mathew MS, Okeke D, Nardi M, Kardys J, Arheart KL. Longitudinal Impact of a Park-Based Afterschool Healthy Weight Program on Modifiable Cardiovascular Disease Risk Factors in Youth. J Community Health. 2018 Feb;43(1):103-116. doi: 10.1007/s10900-017-0393-9. PMID 28689339
- [Background] Messiah SE, D'Agostino EM, Patel HH, Hansen E, Mathew MS, Arheart KL. Sex differences in fitness outcomes among minority youth after participation in a park-based after-school program. Ann Epidemiol. 2018 Jul;28(7):432-439. doi: 10.1016/j.annepidem.2018.03.020. Epub 2018 Apr 12. PMID 29703522
- [Background] D'Agostino EM, Patel HH, Ahmed Z, Hansen E, Sunil Mathew M, Nardi MI, Messiah SE. Impact of change in neighborhood racial/ethnic segregation on cardiovascular health in minority youth attending a park-based afterschool program. Soc Sci Med. 2018 May;205:116-129. doi: 10.1016/j.socscimed.2018.03.038. Epub 2018 Mar 27. PMID 29705630
- [Background] Zewdie H, Zhao AY, Patel HH, Hansen E, Messiah SE, Armstrong SC, Skinner AC, Neshteruk CD, Hipp JA, D'Agostino EM. The association between neighborhood quality, youth physical fitness, and modifiable cardiovascular disease risk factors. Ann Epidemiol. 2021 May;57:30-39. doi: 10.1016/j.annepidem.2021.02.004. Epub 2021 Feb 14. PMID 33596444
- [Background] D'Agostino EM, Patel HH, Hansen E, Mathew MS, Messiah SE. Longitudinal Effects of Transportation Vulnerability on the Association Between Racial/Ethnic Segregation and Youth Cardiovascular Health. J Racial Ethn Health Disparities. 2021 Jun;8(3):618-629. doi: 10.1007/s40615-020-00821-8. Epub 2020 Sep 2. PMID 32880096
- [Background] D'Agostino EM, Patel HH, Ahmed Z, Hansen E, Mathew MS, Nardi MI, Messiah SE. Natural experiment examining the longitudinal association between change in residential segregation and youth cardiovascular health across race/ethnicity and gender in the USA. J Epidemiol Community Health. 2018 Jul;72(7):595-604. doi: 10.1136/jech-2018-210592. Epub 2018 May 10. PMID 29748417
- [Background] D'Agostino EM, Patel HH, Hansen E, Mathew MS, Nardi MI, Messiah SE. Does transportation vulnerability explain the relationship between changes in exposure to segregation and youth cardiovascular health? Health Place. 2019 May;57:265-276. doi: 10.1016/j.healthplace.2019.04.002. Epub 2019 May 24. PMID 31132717
- [Background] Patel HH, Messiah SE, Hansen E, D'Agostino EM. The relationship between transportation vulnerability, school attendance, and free transportation to an afterschool program for youth. Transportation. 2021 Oct;48(5):2315-33.